CLINICAL TRIAL: NCT00412178
Title: Effect of Mobile Communication With a Cellular Phone With a Glucometer on Glucose Control in Type 2 Diabetic Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CMC
Record Dates: First submitted 2006-12-13; First posted 2006-12-15 (Estimated); Last update posted 2006-12-15 (Estimated); Status verified 2006-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Internet; mobile communication; glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Device: telecommunication based glucose monitoring system

SUMMARY:
Previously we demonstrated the beneficial effects of an Internet-based glucose-monitoring system (IBGMS) in people with type 2 diabetes mellitus. The "Diabetes Phone", a cellular phone with a glucometer integrated in the battery pack, was launched in Korea in 2003. Here we test the short-term effectiveness of the diabetes phone for glucose control and compare it with that of IBGMS.

DETAILED DESCRIPTION:
Various strategies using electronic technologies or educational programs have been proposed to improve the quality and efficiency of care for people with diabetes. In the previous study, we introduced a new bidirectional communication tool for diabetes management termed the Internet-Based Glucose Monitoring System (IBGMS), and demonstrated its short-term and long-term effects on glycemic control in type 2 diabetic patients. Other researchers have also showed the effectiveness of telecommunication between health-care providers and patients for maintaining appropriate blood glucose control. These systems allow patients to send data to doctors, identify specific problems and receive recommendations from health-care providers more frequently and with fewer time and place limitations than at traditional face-to-face outpatient clinics. With the IBGMS, physicians can monitor patients' self-monitored blood glucose data at regular intervals, and patients can communicate with their physicians whenever they have any questions. Although bidirectional interactive communications between physicians and patients can be achieved with the IBGMS, there remain time and place limitations. Patients must connect to the Internet using their personal computer to input their data or questions on the IBGMS, while physicians only visit the website at regular intervals unless they have received questions from patients.

To improve the efficiency of communication, we linked the IBGMS to the short message service (SMS) delivered by cellular phone. The patients sent their data to doctors through the IBGMS and then received the doctors' recommendations about adjustment of drug dosage and other related data on the cellular phone. This system improved the efficiency of communication and patients' satisfaction also slightly increased. However, patients were still limited by place and time when sending questions and blood glucose-monitoring data.

Recently, cellular phones have been developed that can measure blood glucose level and transmit data directly to a web server (Diabetes Phone). The combination of a glucometer with the cellular phone function makes it easier for patients to report their self-monitored blood glucose (SMBG) levels and receive feedback from their doctors. However, it was not known how effective this cellular phone glucose-monitoring system would be for control of blood glucose levels, compared to the IBGMS tested previously. We investigated the effectiveness of the diabetes phone for blood glucose control and compared it with that of the IBGMS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus who were able to operate the Internet and to communicate through a mobile phone using the short message service

Exclusion Criteria:

* Significant disease conditions such as symptomatic heart failure, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels more than twice the normal level, renal disease and creatinine level greater than 1.5 mg/dL.
* Patients were also excluded if they participated in other programs that provided information or education about diabetes management from any Internet websites or by any cellular phones other than ours.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-12; Study Completion 2005-04

PRIMARY OUTCOMES:
HbA1c

SECONDARY OUTCOMES:
Compliance

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Hyoung Cho, Instructor, Study Director — Kangnam St. Mary's Hospital, The Catholic University of Korea
Locations (1):
- Kangnam St. Mary's Hospital, The Catholic University of Korea, Seoul, South Korea